CLINICAL TRIAL: NCT01435265
Title: The Effectiveness of Nurse Education and Its Impact on Treatment Adherence in Subjects With Moderate to Severe Psoriasis Undergoing Treatment With Adalimumab
Brief Title: Nurse Education in Subjects With Psoriasis Undergoing Treatment With Adalimumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00009876
Record Dates: First submitted 2011-09-13; First posted 2011-09-16 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Dermatology; Phase IV; Nurse Education; Adalimumab; Humira
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Nurse Education (Active Comparator): Subjects receive normal nurse education materials provided by their physician.
  Interventions: Behavioral: Standard nurse education
- Additional Nurse Education- (Experimental): Subjects will receive additional nurse education beyond the normal education materials provided by their physician
  Interventions: Behavioral: Standard nurse education; Behavioral: Additional nurse education

INTERVENTIONS:
Behavioral: Standard nurse education — Standard-of-care education from a dermatology nurse on the proper use of adalimumab
Behavioral: Additional nurse education — Additional education from a nurse on the use of adalimumab. This will include discussion of the pre-study evaluation with the subject, design of an Individual Educational Plan based on the pre-study evaluation, and a 30-60 minute educational session with the nurse educator at each study visit. Additional information concerning the benefits of the local support group and National Psoriasis Foundation will be provided. Additional education on self-injection and the opportunity to practice self-injection under the supervision of a nurse will also be provided. Subjects will also receive reminder phone calls to take each scheduled dose.
  Arms: Additional Nurse Education-

SUMMARY:
This is a phase IV randomized, prospective open label study to asses the efficacy of an extended nurse eduction program in improving adherence to the prescribed treatment regimen in the treatment of moderate to severe psoriasis vulgaris.

DETAILED DESCRIPTION:
This is a phase IV randomized, prospective open label study to asses the efficacy of an extended nurse eduction program in improving adherence to the prescribed treatment regimen in the treatment of moderate to severe psoriasis vulgaris. Twenty subjects, male or female, ages 18 and older in good health with moderate to severe chronic plaque type psoriasis for whom adalimumab is indicated according to the adalimumab prescribing information. All subjects must have a negative TB skin test according to prescribing guidelines. Subjects must be starting adalimumab for the first time, prescribed by their physician.

This is an open label trial. All subjects will be receiving adalimumab as prescribed by their physician. Half the group will be randomized to receive the additional nurse education program, the other half will receive the normal education materials provided by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female, 18 years of age or greater, in good health with moderate to severe plaque psoriasis for whom adalimumab is indicated according to the adalimumab prescribing information.
* All subjects must have a negative TB skin test according to prescribing guidelines.
* Subjects must be starting adalimumab for the first time, prescribed by their dermatologist.
* Must give written informed consent.
* Subject must be adult males or non-pregnant , non-lactating females.
* Female subjects of childbearing potential must state that they are using measures to avoid conception through active means including, abstinence, oral contraceptives, intrauterine device, Depo-Provera, Norplant, tubal ligation, or vasectomy of the partner in a monogamous relationship.
* Subjects may not be on concomitant systemic medications for their psoriasis such as methotrexate, acitretin, etretinate, cyclosporine, prednisone ot other biological agents or receiving phototherapy at the baseline visit, but no specific washout of these treatments will be required.
* There is no washout for topical medications. Stable dosing of topical medications may be used throughout the duration of the study.

Exclusion Criteria:

* Subjects who have any skin condition or disease that may require concurrent therapy or may confound the evaluation.
* Subjects who have a history of hypersensitivity to adalimumab or history of hypersensitivity to any of the formulation components will be excluded from the study.
* Female subjects who are not postmenopausal for at least one year, surgically sterile or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
* Current enrollment in any research study involving an investigational drug.
* Serious local infection or systemic infection within the three months prior to the first dose of investigational drug.
* Treatment with another investigational drug within one month prior to study drug administration.
* Concurrent treatment with systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine, etanercept, efalizumab, infliximab or mofetil or other systemic immunosuppressant agents.
* Any active or history of HIV, Hepatitis or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Nurse Education | Additional Nurse Education-
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Nurse Education | Additional Nurse Education- | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.7) | 55.0 (9.3) | 51.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Psoriasis Area Severity Index (PASI-75)
Description: The Psoriasis Area Severity Index measures severity of psoriasis on a 0-6 scale for head, trunk, upper extremities, and lower extremities and amount of erythema, infiltration, and desquamation for each area. An overall score of 0-72 for the whole body is calculated from the observed severity values. Outcomes will be reported in terms of PASI 75, or number of participants showing at least 75% reduction in PASI score from baseline. Only final PASI 75 will be reported.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: All participants who completed the study.
Measure: Number; unit: participants
Arm/Group | Normal Nurse Education | Additional Nurse Education-
Number analyzed (Participants) | 3 | 4
participants | 1 | 3

2. Primary Outcome: Investigator's Global Assessment (IGA) of Psoriasis
Description: Investigator's Global Assessment (IGA) is rated on a scale of 0 (clear) to 5 (very severe). The outcome measure to be reported is the number of patients who reached a final IGA of 0 (clear) or 1 (almost clear).
Time Frame: 12 months
Population: All participants completing the study.
Measure: Number; unit: participants
Arm/Group | Normal Nurse Education | Additional Nurse Education-
Number analyzed (Participants) | 3 | 3
participants | 0 | 1

3. Secondary Outcome: Adherence to Adalimumab Treatment
Description: Adherence measured by average days between doses used, as measured by a Medication Event Monitoring System (MEMS) cap on the disposal container for used syringes.
Time Frame: Baseline to 12 months
Population: All participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Normal Nurse Education | Additional Nurse Education-
Number analyzed (Participants) | 3 | 4
days | 19.0 (9.8) | 17.7 (12.1)

ADVERSE EVENTS:
Groups:
- Additional Nurse Education: Experimental: Additional Nurse Education- Subjects will receive additional nurse education beyond the normal education materials provided by their physician
Arm/Group | Normal Nurse Education | Additional Nurse Education
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Nurse Education (N=3) | Additional Nurse Education (N=4)
Abdominal Pain (General disorders) | 1 (1) | 0 (0)
Abscess on R lower leg (Infections and infestations) | 1 (1) | 0 (0)
Blurry/Double vision (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Blood sugar (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Elevated transaminases (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fall-Fractured clavicle and great toe (General disorders) | 1 (1) | 0 (0)
Fatty Liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fibroid tumor (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot and Cold Flashes (General disorders) | 1 (1) | 0 (0)
Increased forehead wrinkling and perioral pigment changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intestinal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mild Hepatic Steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Orthostatic Hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain in L lower back radiating to L leg (muscle strain per PCP) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Possible Keratocanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psoriatic arthritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Severe Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus Infection (General disorders) | 1 (1) | 0 (0)
Sinus drainage (General disorders) | 1 (1) | 0 (0)
Thickening of Cervical Lining (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vaginal yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Worsening of alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
coryza (Infections and infestations) | 0 (0) | 1 (1)
excessive drowsiness/sleepiness (General disorders) | 0 (0) | 1 (1)
recurrent squamous cell carcinoma on R ventral forearm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (2)
Abscess on L side (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — hospitalization for mental abuse from spouse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No